CLINICAL TRIAL: NCT07038655
Title: Investigating the Digestibility, Bioavailability and Utilisation of Varied Combined Protein Sources in Older Males Using a Dual Stable Isotope Tracer Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Philip Atherton, Professor Philip Atherton, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DBU2- FMHS 116-1120
Record Dates: First submitted 2025-05-30; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Healthy Male Volunteers Over 65
Keywords: Digestibility; Muscle Mass; Sarcopenia; Nutrition; Protein
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Drink A (Experimental): 51: 49, casein: soy blend
  Interventions: Dietary Supplement: Randomised 20g Protein Supplement
- Drink B (Experimental): 35: 25: 20: 20, whey: casein: soy: pea blend
  Interventions: Dietary Supplement: Randomised 20g Protein Supplement
- Drink C (Experimental): 35: 25: 20: 20, whey: casein: soy: pea blend
  Interventions: Dietary Supplement: Randomised 20g Protein Supplement
- Drink D (Experimental): 80: 20, casein: whey blend
  Interventions: Dietary Supplement: Randomised 20g Protein Supplement

INTERVENTIONS:
Dietary Supplement: Randomised 20g Protein Supplement — Participants receive a 20g protein feed of their randomised blend over the course of five hours split into aliquots every twenty minutes. The drink also contains a top up of 13C2 leucine stable isotope tracer, as well as uniformly labelled 13C spirulina and 2H labelled free amino acids for quantification of digestibility.

SUMMARY:
By 2020, over 20% of the UK population will be over 65 years of age, dramatically increasing pressure on health and social care. Muscle mass is a strong predictor of healthy ageing and longevity. However, ageing is associated with a progressive loss of muscle, so-called sarcopenia, and this begins in mid-life. Because of the associated loss of muscle strength and stamina, sarcopenia is a major cause of disability, frailty and loss of independence, and is associated with an increased risk of falling and fractures in older people. Strategies to prevent or reduce sarcopenia are receiving increasing attention due to the growing numbers of elderly members of society, but the links between cause and effect are not easy to discern. The investigator's previous work has shown that there are deficits in mechanisms of muscle protein synthesis (MPS) in older people, but why these deficits exist and how they might be countered is still unknown. One of the major problems with ageing is that stimuli which would normally, in younger people, help maintain muscle by turning on MPS (to build muscle) are less effective in older people. The investigator's research has shown that in muscle, the major stimulant of adult human MPS is the availability of the so-called essential amino acids (AA) (which we have to obtain from our diet). After normal feeding, AA and insulin availability both rise, causing net gain of muscle protein. Although these processes do occur in the muscle of older people, they do not occur to the same extent as in the young. Similar results have also been obtained by others, and this is called "anabolic resistance". To exemplify, recent data the investigators have produced showed that: i) increasing the amount of protein provided has a smaller anabolic effect on MPS in older people, and ii) the anabolic response to acute resistance exercise is also less in older people.

Understanding the basic mechanisms underlying age-associated muscle loss would help to define possible counter-measures, such as optimal nutritional strategies. The investigators believe that one contributing factor to the observed "anabolic resistance" of age could be changes in digestive capacity with advancing age, limiting the availability and uptake of ingested dietary proteins. Much of the work to-date relating to protein nutrition and ageing muscle has focussed on whey (WP) and casein proteins (CP), with a wealth of knowledge about the bio-availability of these protein sources across the lifespan. Much less is known about the 'digestibility' of other protein sources (e.g. soy, collagen), with particularly limited knowledge about the interaction between these other protein sources and the second major anabolic stimulus (other than AA feeding), that of resistance exercise. Discovery of a protein blend (PB) with equal capacity for increasing MPS (vs. WP and/or CP)), both at rest and in combination with resistance exercise, plus further knowledge about the bio-availability of different protein sources, will offer new insight for the development of optimal feeding strategies for older adults to counter sarcopenia and the associated health detriments.

In light of difficulties in ileal sampling in studies assessing protein digestibility and absorption in humans, a dual stable isotope approach has been proposed as the ideal solution to determine protein digestibility and absorption; this has been successfully applied and validated in adult humans. This non-invasive approach involves the ingestion of an intrinsically stable isotopically labelled protein, as a single bolus (like a meal) or as intermittent small boluses. Simultaneously, known amounts of differently stable isotopically labelled free amino acids are given with each bolus. The labelled free amino acids are assumed to represent fully digested protein AA and their availability is set at 100, the subsequent appearance of labelled amino acid from the intrinsically labelled protein, of known AA composition and labelling, provides a measure of the digestibility of the protein, as a fraction/percentage of the free AA. In the absence of a suitable intrinsically labelled protein e.g. whey or similar, universally labelled Spirulina (U-13C AA, Cambridge Isotope Laboratories, MA, USA), can be added as a 'labelled or test' protein to any protein meal/source, and report on the digestion of the protein under investigation. This approach has also been successfully applied in patients with cystic fibrosis revealing their reduced ability to digest protein and the positive impact of providing pancreatic enzymes to increase digestion and South Indian children with stunted growth to investigate the digestibility of alternative protein sources i.e. legumes. The investigators aim to use this approach to determine the digestibility of the protein sources in these studies, to assess the bioavailability of amino acids and, in addition, their subsequent utilisation for muscle protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* A BMI <18 or >32 kg·m-2
* Active cardiovascular disease: uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt or recent cardiac event
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial)
* Respiratory disease including pulmonary hypertension or COPD
* Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, types 1 or 2 diabetes (treated and untreated), inborn/ congenital errors of metabolism (e.g. PKU, galactosaemia)
* Active inflammatory bowel disease
* Acute infection
* Acute or chronic renal disease
* Malignancy (or history of malignancy with 5 y)
* Recent steroid treatment (within 6 mo), or hormone replacement therapy
* Coagulopathy
* Musculoskeletal or neurological disorders
* Known allergies to any of the product ingredients

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | Following enrolment, the study period lasts for a single, approximately ten hour day.
  We measure muscle protein synthesis based on the incorporation of 13C2 leucine into the muscle, which is provided through a constant intravenous infusion throughout the study.
Protein Digestibility | Following enrolment, the participants complete a single, approximately ten hour study visit.
  We are measuring the protein digestibility using a dual stable isotope tracer technique. This involves the inclusion of a 13C labelled spirulina protein in the drink alongside a 2H labelled free amino acid mixture. The free amino acid mixture acts as a reference, representing 100% (or complete) digestibility. The spirulina protein acts as a labelled reporter protein, and based on the dilution of the 13C label from this spirulina, we can quantify the digestibility of the experimental protein blends.

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Atherton, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital Medical School, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox J, Phillips BE, Bunce J, Smart T, Wall J, Crossland H, Wilkinson DJ, Smith K, Atherton PJ. Investigating the Digestibility, Bioavailability and Utilization of Protein Blends in Older Adults Using a Dual Stable Isotope Tracer Technique. Nutrients. 2025 Oct 23;17(21):3328. doi: 10.3390/nu17213328. PMID 41228401